CLINICAL TRIAL: NCT02432638
Title: Pierre Robin Sequence Outcome Assessment Multi Institutional Study (PROMIS)
Brief Title: Pierre Robin Sequence Outcome Assessment Multi Institutional Study
Acronym: PROMIS
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution prior to enrollment of subjects
Sponsor: NYU Langone Health (Other)
Collaborators: Indiana University (Other); University of Texas (Other); University of California, Los Angeles (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01966
Record Dates: First submitted 2015-04-10; First posted 2015-05-04 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Pierre Robin Sequence
MeSH Terms: conditions — Pierre Robin Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective, multi-center, longitudinal study is to assess clinical outcomes related to the surgical treatment of PRS ( Pierre Robin Sequence) by MDO (Mandibular distraction osteogenesis). This study aims to develop a scoring system to determine success and complication rate pre and post MDO.

DETAILED DESCRIPTION:
The recruitment phase of this trial is 3 years. Duration of the trial is 19 years.

All study patients who undergo mandibular distraction will be indicated for surgery following published and accepted protocols of care for mandibular distraction in this specific patient population. There will be no experimental/treatment arms in this study. All patients will undergo standard of care interventions and assessments that would not change if the patient were not to participate in this study. The purpose of this study is to follow multiple surgical outcomes following these standard of care practices. The methods and procedures detailed below follow published and accepted standards of care.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent/Assent Form
2. All patients with PRS as defined by mandibular hypoplasia, glossoptosis causing airway obstruction, who undergo MDO prior to the age of 6 months, will be included in the study. This will include all infants regardless of syndromic diagnosis, other organ system abnormalities, cleft palate diagnosis or the presence of other concurrent craniofacial anomalies.

Exclusion Criteria:

1. Infants over the age of 6 months
2. patients who undergo mandibular distraction for conditions other than Pierre Robin sequence.
3. Patient who refuse to be included in this study

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will include all infants under the age of 6 months who undergo mandibular distraction. We will include all racial and ethnic groups as well as both genders. We will not include patients over the age of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Development of Functionality over time | Q 6 years
  We will monitor changes in maxillofacial development, functionality and surgical complications

SECONDARY OUTCOMES:
Cleft Palate Repair outcome | 1 year
  Incidence of airway complications, Incidence of fistula and fistula location

OTHER OUTCOMES:
mandibular growth | 6 years
  as measired by PE, panorex and lateral cephalogram
Long term outcome | 12 and 18 years
  change in AHI or additional airway surgery, incidence of TMJ, tooth development, sensation, scar quality, limitation in jaw excursion

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Flores, MD, Study Chair — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Rachmiel A, Emodi O, Rachmiel D, Aizenbud D. Internal mandibular distraction to relieve airway obstruction in children with severe micrognathia. Int J Oral Maxillofac Surg. 2014 Oct;43(10):1176-81. doi: 10.1016/j.ijom.2014.06.013. Epub 2014 Jul 19. PMID 25052572
- [Background] Runyan CM, Uribe-Rivera A, Karlea A, Meinzen-Derr J, Rothchild D, Saal H, Hopkin RJ, Gordon CB. Cost analysis of mandibular distraction versus tracheostomy in neonates with Pierre Robin sequence. Otolaryngol Head Neck Surg. 2014 Nov;151(5):811-8. doi: 10.1177/0194599814542759. Epub 2014 Jul 22. PMID 25052512
- [Background] Cladis F, Kumar A, Grunwaldt L, Otteson T, Ford M, Losee JE. Pierre Robin Sequence: a perioperative review. Anesth Analg. 2014 Aug;119(2):400-412. doi: 10.1213/ANE.0000000000000301. PMID 25046788
- [Background] Scott AR, Mader NS. Regional variations in the presentation and surgical management of Pierre Robin sequence. Laryngoscope. 2014 Dec;124(12):2818-25. doi: 10.1002/lary.24782. Epub 2014 Jun 26. PMID 24965828
- [Background] Denny AD. Discussion: The surgical correction of Pierre Robin sequence: mandibular distraction osteogenesis versus tongue-lip adhesion. Plast Reconstr Surg. 2014 Jun;133(6):1443-1444. doi: 10.1097/PRS.0000000000000182. No abstract available. PMID 24867726
- [Background] Lee JC, Bradley JP. Surgical considerations in pierre robin sequence. Clin Plast Surg. 2014 Apr;41(2):211-7. doi: 10.1016/j.cps.2013.12.007. Epub 2014 Feb 7. PMID 24607189
- [Background] Murage KP, Tholpady SS, Friel M, Havlik RJ, Flores RL. Outcomes analysis of mandibular distraction osteogenesis for the treatment of Pierre Robin sequence. Plast Reconstr Surg. 2013 Aug;132(2):419-421. doi: 10.1097/PRS.0b013e3182958a54. PMID 23897339
- [Background] Tahiri Y, Viezel-Mathieu A, Aldekhayel S, Lee J, Gilardino M. The effectiveness of mandibular distraction in improving airway obstruction in the pediatric population. Plast Reconstr Surg. 2014 Mar;133(3):352e-359e. doi: 10.1097/01.prs.0000438049.29258.a8. PMID 24572880
- [Background] Paes EC, Fouche JJ, Muradin MS, Speleman L, Kon M, Breugem CC. Tracheostomy versus mandibular distraction osteogenesis in infants with Robin sequence: a comparative cost analysis. Br J Oral Maxillofac Surg. 2014 Mar;52(3):223-9. doi: 10.1016/j.bjoms.2013.11.017. Epub 2013 Dec 30. PMID 24388657
- [Background] Balaraman K, Shanmugakrishnan RR, Bharathi RR, Sabapathy SR. Mandibular distraction in a 75-day-old child with severe Pierre Robin sequence. Indian J Plast Surg. 2013 Jan;46(1):154-6. doi: 10.4103/0970-0358.113743. No abstract available. PMID 23960331
- [Background] Lam DJ, Tabangin ME, Shikary TA, Uribe-Rivera A, Meinzen-Derr JK, de Alarcon A, Billmire DA, Gordon CB. Outcomes of mandibular distraction osteogenesis in the treatment of severe micrognathia. JAMA Otolaryngol Head Neck Surg. 2014 Apr;140(4):338-45. doi: 10.1001/jamaoto.2014.16. PMID 24577483
- [Background] Collins B, Powitzky R, Robledo C, Rose C, Glade R. Airway management in pierre robin sequence: patterns of practice. Cleft Palate Craniofac J. 2014 May;51(3):283-9. doi: 10.1597/12-214. Epub 2013 Jul 22. PMID 23875767
- [Background] Schoemann MB, Burstein FD, Bakthavachalam S, Williams JK. Immediate mandibular distraction in mandibular hypoplasia and upper airway obstruction. J Craniofac Surg. 2012 Nov;23(7 Suppl 1):1981-4. doi: 10.1097/SCS.0b013e31825a64d9. PMID 23154361
- [Background] Cicchetti R, Cascone P, Caresta E, Papoff P, Miano S, Cerasaro C, Ramieri V, Midulla F, Moretti C. Mandibular distraction osteogenesis for neonates with Pierre Robin sequence and airway obstruction. J Matern Fetal Neonatal Med. 2012 Oct;25 Suppl 4:141-3. doi: 10.3109/14767058.2012.715011. PMID 22958047
- [Background] Scott AR, Tibesar RJ, Sidman JD. Pierre Robin Sequence: evaluation, management, indications for surgery, and pitfalls. Otolaryngol Clin North Am. 2012 Jun;45(3):695-710, ix. doi: 10.1016/j.otc.2012.03.007. PMID 22588044
- [Background] Sesenna E, Magri AS, Magnani C, Brevi BC, Anghinoni ML. Mandibular distraction in neonates: indications, technique, results. Ital J Pediatr. 2012 Feb 2;38:7. doi: 10.1186/1824-7288-38-7. PMID 22300418